CLINICAL TRIAL: NCT01305460
Title: A Phase I/II Study of the Efficacy and Safety of an Intensified Schedule of Azacitidine (Vidaza®) in Intermediate-2 and High Risk MDS Patients
Brief Title: Intensified Azacitidine in High Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-AZA intensif
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine intensified dose (Experimental)
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Treatment will consist of azacitidine 75mg/m2/d for 5 days every 14 days for 4 cycles.
  * Patients achieving CR or PR will be then treated with 4 cycles of azacitidine 75mg/m2/d for 5 days every 21 days followed by cycles of azacitidine 75mg/m2/d for 7 days administered every 28 days (cycles 9 and beyond), to be continued until progression/relapse or toxicity arises.
  * Patients not obtaining CR or PR after the initial 4 cycles of azacitidine-14 will continue to receive azacitidine 75mg/m2/d for 5 days every 14 days for 4 additional cycles (cycles 5 to 8). If they achieve CR, PR or HI after 8 cycles, they will then be treated with azacitidine 75mg/m2/d for 5 days every 21 days (cycles 9 to 12) and subsequently cycles of azacitidine 75mg/m2/d for 7 days administered every 28 days (cycles 13 and beyond) until progression/relapse or toxicity arises.
  * Patients not obtaining CR, PR or HI after 8 cycles of azacitidine-14 will go "off-study".
  Other Names: Vidaza

SUMMARY:
A phase I/II study of the efficacy and safety of an intensified schedule of Azacitidine (Vidaza®) in intermediate-2 and high risk MDS patients.

DETAILED DESCRIPTION:
The study is an open-label, multicenter phase I/II study.

Treatment Regimen, Dosage and Duration:

Treatment will consist of azacitidine 75mg/m2/d for 5 days every 14 days for 4 cycles (azacitidine-14, cycles 1-4).

* Patients achieving CR or PR will be then treated with 4 cycles of azacitidine 75mg/m2/d for 5 days administered every 21 days (azacitidine-21, cycles 5 to 8) followed by cycles of azacitidine 75mg/m2/d for 7 days administered every 28 days (azacitidine-28, cycles 9 and beyond), to be continued until progression/relapse or toxicity arises).
* Patients not obtaining CR or PR after the initial 4 cycles of azacitidine-14 will continue to receive azacitidine 75mg/m2/d for 5 days every 14 days for 4 additional cycles (cycles 5 to 8). If they achieve CR, PR or HI after 8 cycles, they will then be treated with azacitidine 75mg/m2/d for 5 days every 21 days (azacitidine-21, cycles 9 to 12) and subsequently cycles of azacitidine 75mg/m2/d for 7 days administered every 28 days (azacitidine-28, cycles 13 and beyond) until progression/relapse or toxicity arises.
* Patients not obtaining CR, PR or HI after 8 cycles of azacitidine-14 will go "off-study".

Number of patients to be included:

The trial will enroll at least 27 patients (phase I of the trial) and a maximum of 81 patients (phase II of the trial). A safety analysis will be performed by an independent DSMB after inclusion of 9, 18 and 27 patients. This safety analysis will focus particularly on the clinical consequences of cytopenias. Moreover, a teleconference will be organized twice monthly between the PI and investigators to share safety observations and take appropriate actions if needed. CRFs will be collected every cycle focusing particularly on the safety of this dose intensified study. All AE and SAE will be reported to the DSMB upon reception.

Primary Endpoint:

-Response rate (including CR and PR) according to IWG 2006 criteria for MDS after 4 and 8 cycles 75mg/m2/d azacitidine administered every 2 weeks.

Secondary Endpoints:

* Safety/toxicity profile of azacitidine administered every 14 days (NCI-CTAE)
* Responses (CR, PR, marrow CR, HI) according to IWG 2006 criteria and their duration
* Overall survival and progression (IPSS/AML) free survival.

Sample Size and Duration of Trial:

The first stage of the trial will include 27 patients. The trial will be terminated if 9 or fewer responses are observed. Otherwise, additional patients will be recruited in the second stage until a total sample size of 81 patients is reached.

Duration of inclusion: 24 months for 81 patients Duration of follow-up: 24 months

ELIGIBILITY:
Inclusion Criteria:

* MDS defined according to WHO classification (also including RAEB-T according to FAB classification) (see appendix 1) with intermediate-2 or high risk IPSS (see appendix 1).
* Age ≥ 18 years and <75 years.
* Must understand and voluntarily sign an informed consent form.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Patients must have ECOG performance status (PS) of 0 - 2, and no major comorbidities preventing administration of an intensified regimen of azacitidine.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must :
* Have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study. Lactating patients are excluded.
* Agree to use, and to be able to comply with, effective contraception without interruption, 4 weeks before starting study drug throughout the entire duration study drug therapy (including doses interruptions) and for 3 months after the end of the study drug therapy.
* Male patients must :
* Agree the need for the use of a condom if engaged in sexual activity with a woman of childbearing potential during the entire period of treatment, even if disruption of treatment and during 3 months after end of treatment.
* Agree to learn about the procedures for preservation of sperm before starting treatment.
* Creatinine < 1.5 N or estimated clearance of creatinine above 30 ml/min.
* Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) < 3.0 x upper limit of normal (ULN).
* Serum total bilirubin < 1.5 mg/dL. (except for unconjugated hyperbilirubinemia due to Gilbert's disease or secondary to MDS-related dyserythropoiesis).
* Health insurance

Exclusion Criteria:

* Patients with a history of myeloproliferative syndrome or CMML.
* Known positive status for human immunodeficiency virus (HIV) or hepatitis B or C.
* Pregnant and lactating patients are excluded because the effects of azacitidine on a fetus or a breast-fed child are unknown.
* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection, symptomatic congestive heart failure (NYHA > II), cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients receiving any other standard or investigational cytotoxic treatment for their hematologic malignancy in the last 8 weeks
* Any medical condition which in the opinion of the investigator places the patient at an unacceptably high risk for toxicities of an intensified regimen of azacitidine.
* Less than 6 months since prior allogeneic bone marrow transplantation.
* Less than 3 months since prior autologous bone marrow or stem cell transplantation
* Active cancer or prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 3 years.
* Prior treatment with azacitidine.
* Known allergy/intolerance to azacitidine or mannitol.
* ECOG > 2.
* Life expectancy of less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-07-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2015-11-16 (Actual)

PRIMARY OUTCOMES:
Response rate (including CR and PR) according to IWG 2006 criteria for MDS after 4 and 8 cycles 75mg/m2/d azacitidine administered every 2 weeks. | 2 months
  After 4 courses treatment

SECONDARY OUTCOMES:
Safety/toxicity profile of azacitidine administered every 14 days (NCI-CTAE) | 1-24 months
  After each course of treatment until end of treatment.
Responses (CR, PR, marrow CR, HI) according to IWG 2006 criteria and their duration. | 2-4 months
  After 4 and 8 courses of treatment.
Overall survival and progression (IPSS/AML) free survival. | 2 months and further
  After 4 course of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Adès, MD, Study Chair — Groupe Francophone des Myélodysplasies; Simone Boehrer, MD, Principal Investigator — Groupe Francophone des Myélodysplasies
Locations (21):
- France (21):
  - CHU d'Amiens, Amiens
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - Centre henri Mondor, Créteil
  - CHU Albert Michallon - Service d'Hématologie Clinique, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - Hôpital Huriez, Lille
  - Hôpital Paoli Calmettes, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - CHU Brabois, Nancy
  - CHU de nantes, Nantes
  - Hôpital l'Archet de Nice, Nice
  - Hôpital Cochin, Paris
  - Hôpital Saint Louis, Paris
  - Hopital Saint Louis - AP-HP, Hematology Dpt, Paris
  - CHU de Haut-Lévèque, Pessac
  - CHU de Poitiers, Poitiers
  - CHRU Annecy Hospital, Pringy
  - Hôpital Pontchaillou, Rennes
  - Hopital Purpan Service d'Hématologie Clinique, Toulouse
  - CH de Valence, Valence

REFERENCES:
- See also: Website of the Groupe Francophone des Myélodysplasies (GFM) — http://www.gfmgroup.org